CLINICAL TRIAL: NCT05439291
Title: Comparing Operative vs Non Operative Treatment for Pilonidal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Bill Chiu, MD, Associate Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-65058
Record Dates: First submitted 2022-06-09; First posted 2022-06-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pilonidal Disease
Keywords: Pilonidal Surgery; Pilonidal Excision; Pilonidal recurrence

STUDY DESIGN:
Intervention Model Description: The research will consist of randomized 1:1 controlled trial comparing regular epilation regimen only vs. regular epilation regimen with surgical excision
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular epilation regimen only (Active Comparator)
  Interventions: Procedure: Regular Epilation Regimen
- Regular epilation regimen with surgical excision (Active Comparator)
  Interventions: Procedure: Regular Epilation Regimen; Procedure: Surgical excision

INTERVENTIONS:
Procedure: Regular Epilation Regimen — Epilation using laser device
Procedure: Surgical excision — Excision of pilonidal pit with trephine
  Arms: Regular epilation regimen with surgical excision

SUMMARY:
The goal is to evaluate whether surgical excision of the pilonidal disease is needed after resolution of the initial symptoms when the patient follows regular hair removal regimen such as laser epilation.

DETAILED DESCRIPTION:
The goal is to evaluate whether surgical excision of the pilonidal disease is needed after resolution of the initial symptoms when the patient follows regular hair removal regimen such as laser epilation. Patients with pilonidal disease can have significant pain and drainage at the gluteal cleft, and recurrent disease in this teenage and young adult population often leads to social embarrassment, isolation, and time off from work or school. Effective therapy to prevent recurrent disease is urgently needed.

The current standard of care is excision of pilonidal cyst. The research will consist of randomized 1:1 controlled trial comparing regular epilation regimen only vs. regular epilation regimen with surgical excision. The research will consist of patient surveys and clinical notes. Surgical excision is not needed to be part of this research.

All patients will receive surveys and their charts will be reviewed. At the point of treatment decision making, the patients will be randomized to one of the two options.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Stanford Healthcare with pilonidal disease.
* Patients over the age of 8yrs.

Exclusion Criteria:

* Inability to read, write or understand English ***or Spanish
* Intellectual disability precluding the patient from being able to comprehend or respond to the questionnaire

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrent symptoms of pilonidal disease | Up to 1 year

SECONDARY OUTCOMES:
Number of participants requiring antibiotic treatment | Up to 1 year
Time taken off from school or work due to pilonidal disease | Up to 1 year
Effect on parent's daily activities | Baseline to 1 year
  Parents measure the effect of caring for afflicted children on a 0-10 rating scale, higher scores correspond to more difficulties.
Number of participants requiring additional surgical intervention | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bill Chiu, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No